CLINICAL TRIAL: NCT03974659
Title: Through the Navigation Transcranial Magnetic Stimulation Over the Language Key Areas of Cerebellar to Enhance Language Function Recovery After Brain Tumor Resection
Brief Title: Enhanced Recovery After Surgery Using TMS on Cerebellar Language Area for Brain Tumor Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Jing'an Central Hospital (Unknown); Huashan Hospital North Hospital (Unknown)
Responsible Party: Principal Investigator, Jinsong Wu, Principal Investigator, Clinical Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY2018-395
Record Dates: First submitted 2019-05-20; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-10

CONDITIONS: Cerebellar Function; Transcranial Magnetic Stimulation; Language Disorders
MeSH Terms: conditions — Language Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: A Prospective Randomized, Double-Blind Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Theta Burst Stimulation (Active Comparator): Intervention group: ten consecutive days bilateral cerebellar VIIa lobules Theta Burst Stimulation.
  Intermittent Theta Burst Stimulation(Positive stimulation) is used in right cerebellar VIIa lobule.Each stimulus had three 50 Hz monopulses, which were repeated every 200 ms. Each stimulation continued for 2 seconds and rested for 8 seconds. The total intervention time was 200s (600 pulses) Continuous Theta Burst Stimulation(Negative stimulation) is used in left cerebellar VIIa lobule,three 50 Hz monopulses in each stimulus, each with an interval of 200 ms, and each intervention lasted 40s (600 pulses).
  The stimulation intensity was 80% Rest Motor Threshold.According to the patients' condition, age and tolerance,the intensity should be adjusted.
  Interventions: Combination Product: Transcranial magnetic stimulation
- sham Theta Burst Stimulation (Sham Comparator): sham group: we flip coil to make fake stimulation, the stimulation will also make sounds, but no magnetic field effect, the stimulation mode is the same as the intervention group.
  Interventions: Combination Product: Transcranial magnetic stimulation

INTERVENTIONS:
Combination Product: Transcranial magnetic stimulation — 1.Patients were given 10 consecutive days bilateral cerebellar VIIa lobules Theta Burst Stimulation which was a special mode of Transcranial magnetic stimulation from one week after surgery Intermittent Theta Burst Stimulation(Positive stimulation) is used in right cerebellar VIIa lobule.Each stimulus had three 50 Hz monopulses, which were repeated every 200 ms. Each stimulation continued for 2 seconds and rested for 8 seconds. The total intervention time was 200s (600 pulses) Continuous Theta Burst Stimulation(Negative stimulation) is used in left cerebellar VIIa lobule,three 50 Hz monopulses in each stimulus, each with an interval of 200 ms, and each intervention lasted 40s (600 pulses).
  Other Names: speech rehabilitation training

SUMMARY:
At present, the incidence of language dysfunction in patients with brain language area tumor in the first month after operation was 20%-40%. The investigator's team has confirmed and found that bilateral cerebellar VIIa lobules are the critical areas of cerebellar which is closely related to the language function of the patients. This study aims at enhancing language function recovery after surgery through the transcranial magnetic stimulation stimulates the key areas of cerebellar.

This study is a prospective, randomized, double-blind, multi-center clinical trial in which participants with postoperative aphasia in the brain-language region tumors of three neurosurgery departments, Huashan Hospital, Shanghai Jing'an Center Hospital and Huashan Hospital North Hospital. Participants were randomly divided into Intervention group and control group. Before transcranial magnetic stimulation treatment, the two groups were required to conduct language behavior assessment and magnetic resonance imaging data. Participants in both groups were given 10 consecutive days bilateral cerebellar VIIa lobules Theta Burst Stimulation from one week after surgery and received speech rehabilitation training after stimulation.

The investigators collect patients MRI data and language behavioral assessment scores at 1week post operation and 1 month after the operation and 3 months after the operation. Subsequently, three MRI data and language behavioral assessment scores were processed and statistically analyzed to compare the differences between the two groups

DETAILED DESCRIPTION:
Intervention group: Intermittent Theta Burst Stimulation(Positive stimulation) is used in right cerebellar VIIa lobule. Continuous Theta Burst Stimulation(Negative stimulation) is used in left cerebellar VIIa lobule. The stimulation intensity was 80% Rest Motor Threshold.According to the patients' condition, age and tolerance,the intensity should be adjusted.

Control group: The investigators use with fake stimulation , the appearance is the same as the magnetic stimulator used in the experimental group, and the stimulation will also make sounds, but no magnetic field effect, the stimulation mode is the same as the intervention group.

Subsequently, The investigators collect patients MRI data and language behavioral assessment scores at 1week post operation and 1 month after the operation and 3 months after the operation.three times MRI data and language behavioral assessment scores were processed and statistically analyzed to compare the differences between the two groups from the cerebellar spontaneous neurological activity level (ALFF), cerebellar gray matter volume, functional connectivity of cerebellar network and language behavioral score.

ELIGIBILITY:
Inclusion Criteria:

* Language dysfunction after brain tumor surgery (aphasia quotient,AQ)< 93.8
* Chinese mother tongue
* Right handedness confirmed by Edinburgh Handedness Scale
* Tumor patients with linguistic region involvement in the dominant hemisphere
* Karnofsky Performance Status (KPS)< 70
* Voluntary participation in this project

Exclusion Criteria:

* Patients with frequent epileptic seizures (> 2 epilepsy episodes per week)
* Previous implants of metal pacemakers, stimulators, hearing aids, dentures, and insulin pumps or claustrophobia
* People with a history of psychiatric disorders
* Patients with severe medical diseases
* Patients with Alzheimer's disease and Parkinson's disease. Medical diseases
* Pregnant women
* Other clinical trials in the same period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Boston naming test | Change from postoperative 1 week to postoperative 1month & postoperative 3 months
  The change of Boston naming test scores is being assessed
MMSE | Change from postoperative 1 week to postoperative 1month & postoperative 3 months
  The change of Mini-mental State Examination scores is being assessed
ABC | Change from postoperative 1 week to postoperative 1month & postoperative 3 months
  Aphasia Battery of Chinese，Conclude naming, repeating, comprehend and spontaneous speech test，The change of ABC scores is being assessed
ALFF | Change from postoperative 1 week to postoperative 1month & postoperative 3 months
  The change of Cerebellar spontaneous neurological activity level is being assessed
Cerebellar gray matter volume | Change from postoperative 1 week to postoperative 1month & postoperative 3 months
  The change of Cerebellar gray matter volume is being assessed
Functional connectivity of cerebellar network | Change from postoperative 1 week to postoperative 1month & postoperative 3 months
  The change of functional connectivity of cerebellar network is being assessed

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, MD, Principal Investigator — Huashan Hospital
Locations (2):
- China (2):
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Jing'an Central Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No